CLINICAL TRIAL: NCT00130286
Title: Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Recombinant Human Growth Hormone and/or Rosiglitazone in the Treatment of Human Immunodeficiency Virus-Associated Visceral Adiposity and Insulin Resistance
Brief Title: Growth Hormone and/or Rosiglitazone for HIV-Associated Increased Abdominal Fat and Insulin Resistance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marshall Jay Glesby, MD, PhD, Professor of Medicine and Public Health, Weill Medical College of Cornell University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65515; R01DK065515 (NIH)
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: HIV-Associated Lipodystrophy Syndrome; Insulin Resistance; HIV Infections; Metabolic Syndrome X; Body Weight Changes
Keywords: Lipodystrophy; HIV; Growth hormone; Rosiglitazone; Visceral fat; Metabolic syndrome; Treatment Experienced; Visceral fat accumulation; fat accumulation; HIV-Associated Metabolic Syndrome
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Insulin Resistance; HIV Infections; Metabolic Syndrome; Body Weight Changes; Lipodystrophy | interventions — Rosiglitazone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rhGH + rosi (Experimental): Recombinant human growth hormone + rosiglitazone
  Interventions: Drug: Rosiglitazone; Drug: Recombinant human growth hormone + rosiglitazone
- rhGH placebo + rosi (Experimental): Placebo for recombinant human growth hormone + rosiglitazone
  Interventions: Drug: Rosiglitazone; Drug: Recombinant human growth hormone + rosiglitazone
- rhGH + rosi placebo (Experimental): Recombinant human growth hormone + placebo for rosiglitazone
  Interventions: Drug: Rosiglitazone; Drug: Recombinant human growth hormone + rosiglitazone
- Double placebo (Placebo Comparator): Placebo for recombinant human growth hormone + placebo for rosiglitazone
  Interventions: Drug: Rosiglitazone; Drug: Recombinant human growth hormone + rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg tablet twice a day x 12 weeks (double-blind phase)
Drug: Recombinant human growth hormone + rosiglitazone — Recombinant human growth hormone or placebo 3 mg s.c. x 12 weeks (double-blind phase)

SUMMARY:
The purpose of the study is to determine if the combination of recombinant human growth hormone plus rosiglitazone (an insulin-sensitizing drug) is safe and more effective than either drug alone (or no active therapy) for the treatment of fat accumulation in people with HIV infection and insulin resistance.

DETAILED DESCRIPTION:
A number of people with HIV infection who gain weight in the abdomen (sometimes called lipodystrophy) also have a high level of the sugar-controlling hormone called insulin. These people need to produce this extra insulin to help keep their blood sugar normal. This is called "insulin resistance."

Studies have shown that growth hormone (also called "Serostim") can decrease abdominal fat, but it can also worsen the insulin resistance. Rosiglitazone (also called "Avandia") is used to treat insulin resistance in people who have diabetes, so we want to see if taking growth hormone and rosiglitazone together will be better for treating the fat accumulation part of lipodystrophy than either drug alone or no active therapy.

The study is 24 weeks long, divided into two 12-week parts.

The first part of the study is double-blind, meaning that neither participants nor the study staff will know which drugs participants are on. Participants will be assigned randomly (like flipping a coin) to one of four groups:

1. Growth hormone (one injection, daily) PLUS rosiglitazone (one tablet, twice daily).
2. Growth hormone PLUS rosiglitazone placebo ("sugar pill").
3. Growth hormone placebo (plain water injection) PLUS rosiglitazone.
4. Growth hormone placebo PLUS rosiglitazone placebo.

Everyone in the study will need to be hospitalized overnight for special tests at the beginning of the study and at week 12.

The second part of the study is open-label, meaning that participants and the study staff will know which drugs participants are receiving. All volunteers will receive both active drugs:

* Growth hormone (one 2 mg injection, every other day) PLUS rosiglitazone (one 4 mg tablet, twice daily).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* On stable Food and Drug Administration (FDA)-approved antiretrovirals for at least 8 weeks
* Excess abdominal fat based on waist and hip measurements done at the screening visit. [waist greater than 34.7 inches (men) or 29.6 inches (women) and waist to hip ratio greater than 0.95 (men) or 0.9 (women)]
* Evidence of insulin resistance (based on fasting glucose and insulin levels done at screening)
* Triglycerides less than 750 mg/dL

Exclusion Criteria:

* Pregnancy
* Active AIDS-defining infection or other acute illness, within 30 days of entry.
* Active cancer (except for localized Kaposi's sarcoma) or active brain tumor
* Any diagnosis of pancreatitis, carpal tunnel syndrome, diabetes, angina, coronary artery disease, or disorder associated with fluid retention (examples: cirrhosis, congestive heart failure)
* Untreated or uncontrolled high blood pressure, within 30 days of entry.
* Within 12 weeks of study entry, use of the following:

  * Obesity (fat-reducing) drugs.
  * Anti-diabetic or insulin-sensitizing drugs (examples: rosiglitazone, pioglitazone, or metformin).
  * Systemic glucocorticoids (example: prednisone).
  * Growth hormone or any medication for AIDS-associated wasting.
  * Systemic chemotherapy, interferon, or radiation therapy.
  * Androgenic agents [examples: nandrolone, oxandrolone (Oxandrin) (testosterone replacement therapy is permitted if started more than 30 days before entry)]
  * Appetite stimulants (Marinol, Megace, Periactin).
* Use of cholesterol lowering drugs, unless started more than 12 weeks before entry
* Inability to have a magnetic resonance imaging (MRI) scan performed (examples: cardiac pacemaker, intracranial aneurysm clips)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall J Glesby, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - AIDS Community Research Initiative of America (ACRIA), New York, New York
  - Cornell HIV Clinical Trials Unit, Weill Medical College of Cornell University, New York, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - Columbia University College of Physicians and Surgeons, New York, New York

REFERENCES:
- [Result] Glesby MJ, Albu J, Chiu YL, Ham K, Engelson E, He Q, Muthukrishnan V, Ginsberg HN, Donovan D, Ernst J, Lesser M, Kotler DP. Recombinant human growth hormone and rosiglitazone for abdominal fat accumulation in HIV-infected patients with insulin resistance: a randomized, double-blind, placebo-controlled, factorial trial. PLoS One. 2013 Apr 12;8(4):e61160. doi: 10.1371/journal.pone.0061160. Print 2013. PMID 23593417
- [Derived] Kotler DP, He Q, Engelson ES, Albu JB, Glesby MJ. The effect of recombinant human growth hormone with or without rosiglitazone on hepatic fat content in HIV-1-infected individuals: a randomized clinical trial. Antivir Ther. 2016;21(2):107-16. doi: 10.3851/IMP2927. Epub 2014 Dec 23. PMID 25536669

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo
Started | 22 | 19 | 17 | 19
Completed | 22 | 16 | 13 | 17
Not Completed | 0 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Missing lab specimens | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo | Total
Number analyzed (Participants) | 22 | 19 | 17 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.4) | 49.3 (6.1) | 48.6 (4.9) | 46.6 (6.7) | 47.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 6 | 17
  Male | 18 | 15 | 14 | 13 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 6 | 6 | 24
  White | 15 | 11 | 11 | 12 | 49
  More than one race | 1 | 2 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 3 | 9 | 30
  Not Hispanic or Latino | 13 | 10 | 14 | 10 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity
Description: Change in insulin sensitivity value from baseline to week 12 by frequently sampled intravenous glucose tolerance test
  This assessment was only conducted at baseline and week 12; therefore the change reflects the difference between these two time points.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: uU*10^-4*min*ml^-1
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo
Number analyzed (Participants) | 22 | 16 | 13 | 17
uU*10^-4*min*ml^-1 | 0.20 [-0.37 to 1.00] | 1.44 [0.68 to 2.59] | -0.63 [-1.03 to 0.11] | 0.14 [-0.41 to 1.21]

2. Secondary Outcome: Change in Visceral Adipose Tissue Volume
Description: Change in visceral adipose tissue volume from baseline to week 12 measured by whole body MRI
  Data are presented only for subjects who had MRI scans done at both time points.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: L
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo
Number analyzed (Participants) | 20 | 15 | 11 | 16
L | -1.13 (1.41) | -0.19 (0.69) | -1.15 (0.81) | -0.04 (0.9)

3. Secondary Outcome: Change in Subcutaneous Adipose Tissue Volume
Description: Change in subcutaneous adipose tissue volume from baseline to week 12 by whole body MRI
  Data are presented only for subjects who had MRI scans done at both time points.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: L
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo
Number analyzed (Participants) | 20 | 15 | 11 | 16
L | -0.11 (3.33) | 0.74 (1.86) | -0.38 (1.23) | -0.03 (2.64)

ADVERSE EVENTS:
Description: The denominator for adverse events by treatment arm reflects the number of subjects who initiated study treatment in each arm. The denominator for serious adverse events reflects the number of randomized subjects since one serious adverse event occurred in someone who never initiated study drugs. Therefore the denominators differ.
Arm/Group | rhGH + Rosi | rhGH Placebo + Rosi | rhGH + Rosi Placebo | Double Placebo
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/19 | 0/17 | 3/19
Other Adverse Events (participants affected / at risk) | 17/22 | 11/18 | 14/15 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhGH + Rosi (N=22) | rhGH Placebo + Rosi (N=19) | rhGH + Rosi Placebo (N=17) | Double Placebo (N=19)
Delirium (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient with underlying seizure disorder who was nonadherent with anticonvulsant therapy and withdrawing from methadone. The delirium was attributed to a post-ictal state.
Study drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient injected rhGH or placebo twice daily instead of once daily but had no adverse effects. She was ultimately found to be on rhGH placebo.
Fever of undetermined origin (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — FUO was considered not related to study drugs. Ultimately found to be on doube placebo.
Leg weakness and pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient with known myelopathy and multiple episodes of leg pain and weakness was admitted to the hospital with recurrent symptoms thought to be unrelated to study drugs. Ultimately found to be on double placebo.
Ureteral obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient admitted to hospital with ureteral obstruction due to a kidney stone. Had known history of nephrolithiasis. Ultimately found to be on double placebo.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rhGH + Rosi (N=22) | rhGH Placebo + Rosi (N=18) | rhGH + Rosi Placebo (N=15) | Double Placebo (N=17)
Fever (General disorders) | 0 | 1 | 1 | 2
Fatigue (General disorders) | 7 | 6 | 5 | 5
Weight gain (General disorders) | 1 | 0 | 1 | 2
Headache (General disorders) | 3 | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 5 | 5
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6 | 3
Parethesias (Nervous system disorders) | 5 | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Hyperglycemia (Endocrine disorders) | 5 | 1 | 8 | 2
Increased ALT (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Increased AST (Hepatobiliary disorders) | 1 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Edema (Musculoskeletal and connective tissue disorders) | 12 | 3 | 11 | 2
Breast enlargement/tenderness (Reproductive system and breast disorders) | 4 | 1 | 0 | 0
Cough/upper respiratory infection (General disorders) | 0 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No